CLINICAL TRIAL: NCT00677846
Title: Venous Thrombus Investigation With Contrast Enhanced Ultrasound Imaging, a Follow up Study
Brief Title: Venous Thrombus Investigation With Contrast Enhanced Ultrasound Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Prof. Dr. C. Hehrlein, Abteilung Innere Medizin III, Kardiologie u. Angiologie
Other Study IDs: 314/03
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Deep Venous Thrombosis
Keywords: contrast agent ultrasound, vein thrombosis, vascularization
MeSH Terms: conditions — Venous Thrombosis; Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3: Patients with symptoms of deep venous thrombosis less than for 2 weeks, with thrombus occluding without any reperfusion in color mode in the common femoral vein (CFV), the femoral vein (FV) or the popliteal vein (PV)

SUMMARY:
Background:

During the repair process of deep venous thrombosis, capillary formation is seen from day 18 to day 25. Contrast agent investigation is well known to detect small vessels in arterial disease. We intend to use this method to detect early vascularisation in the thrombus, in order to get more information about the evolution of the thrombosis in vivo.

Aims of the study:

Investigation of a newly diagnosed occluding venous thrombus with duplexsonography, using contrast agent and compare the degree of vascularization in the same patient after 3 weeks and 3 months. The relative signal intensity difference (baseline to peak) of the time intensity curve (TIC) is measured in defined region of interests (ROI). Comparison of the visibility of revascularisation between color duplexsonography, power mode and contrast agent will be done.

Method:

Patients with venous thrombosis of the proximal limb veins (femoral or popliteal vein) will be investigated with ultrasound agent in supine position. 5 ml of the contrast agent sulfur hexafluoride is given intravenously into a vein of the dorsal foot. The measurements are done in a defined area, where the thrombus is fully occluding in color Doppler investigation. The regions of interest will be the vessel walls and the centre of the thrombus in cross section view. The signal intensities are measured at baseline and peak (in decibel) in the centre and in the peripheral part of the vein. 20 patients with acute deep venous thrombosis will be included in this pilot study and investigated at baseline, after 3 weeks and 3 months.

Previously (before contrast agent application), the veins are investigated with color - and power Doppler to test visibility in comparison to the contrast agent investigation.

DETAILED DESCRIPTION:
1. Study set up and Study design

   It will be an open, non-randomized prospective clinical pilot study to assess the value of contrast agents in venous thrombus investigations.

   a. Hypothesis
   * The relative signal intensity increase in decibel after intravenous contrast media injection as a tool to measure thrombus - revascularization, assessed in defined regions of interests in the thrombus is smaller in acute occluding (< 2 week) thrombosis compared to the follow up measurements after 3 months in the same patient.
   * Visibility of revascularization is increased with contrast agent compared to color Doppler - and power Doppler investigation assessed by 2 independent investigators
2. Methods

   1. Clinical investigation

      All patients and subjects will be investigated clinically. The patient's family history as well as the present and past history for deep venous thrombosis is assessed. The first day of symptoms of the deep vein thrombosis is noted. The thromboembolic disease is assessed clinically using the Wells' score.

      In addition the pulses of the dorsal foot artery are palpated. Height and weight are assessed as well as medication intake, especially dose and type of anticoagulation therapy. Laboratory testing will include C-reactive protein and D-Dimer test at visit 1, 2 and 3, as well as thrombophilia screening (anti-thrombin, anti protein C resistance, protein C, protein S, Lupus anticoagulans, prothrombinfragment 1 and 2, factor II mutation G 202 10 A)
   2. Duplexsonography investigation

      All patients with proximal deep venous thrombosis are evaluated for study inclusion. The eligible patients are investigated in supine position in both legs with B-mode - compression sonography and Doppler spectral analysis. The vein segments are considered affected if they are incompressible and if no Doppler spectrum is assessable. The most proximal fully occluding thrombus area (in color mode) is defined and the localization is measured in cm from the groin or the popliteal line. The particular area of interest is investigated in cross section with color duplex sonography and power Doppler using the linear wideband scan head L7 (5-12 MHz) of the duplexsonography device GE LOGIC 9 (GE Healthcare Technologies, Ultrasound Milwaukee, WI, USA). One cineloop of 20 seconds each are saved in real time assessment. The sequences are saved in avi - and in dicom - format for each Doppler specification. The saved films will be evaluated offline by two different investigators using a visibility score.

      Duplexsonography investigation with contrast agent:

      Five ml of the contrast agent sulfur hexafluoride (= SonoVueTM, Bracco International B.V., Amsterdam, the Netherlands) is given intravenously into a superficial vein of the dorsal foot or calf of the leg investigated (green butterfly needle 20 gauge). If no leg veins are available the arm vein route will be used. The measurements are done in the fully occluding thrombus area in cross section. The area will be localized in order to find the same point of investigation again at visit 2 and visit 3.

      The following settings are applied in all cases of contrast agent investigations: Contrast program preset with low mechanical index (MI) of < 0.13 (acoustic output 4 %), depth 4 - 5 cm, one focus zone adapted to the depth of the investigated vein area, dynamic range 72, pulse repetition interval 1.25, B (brightness-)-mode amplification 30. The ultrasound pulses will not be triggered. An optimized manual technique is applied to minimize movement artefacts. After 10 seconds of B-mode assessment, a bolus of 5 ml SonoVueTM solution will be injected into a peripheral foot or calf vein using a butterfly needle (20 gauge). The SonoVueTM - injection is followed immediately by 10 ml saline bolus to flush the injection line. The investigations will be documented by digital saving of the cineloops in avi- and dicom format. Image analysis is performed offline, using the time intensity curve (TIC) analysis program provided by GE Healthcare Technologies, implemented into the LOGIQ 9 ultrasound system. Using the ultrasound raw data, the image displays the acoustic intensity measured in decibel (dB) during acquisition time in the manually defined region of interest (ROI) i.e. the vessel wall and the intraluminal thrombus in cross section. The signal intensities are measured at baseline and peak (in decibel) in the centre and in the peripheral part of the vein. The differences are calculated. Measurements are done 3 times, mean values are used for further calculation.

      20 patients with acute deep venous thrombosis with symptom onset within the last 2 weeks will be included in this pilot study. The patients are followed for 3 months, the parameters are assessed and compared intraindividually.
   3. Visibility score

      The three documented investigations of each patient in color - and power Doppler-mode as well as the contrast agent assessment are evaluated by two different blinded persons, experienced in ultrasound investigation (> 2000 ultrasound investigations, specialty degree in ultrasound investigation IP and DG). The visibility score according to the one described by Gehrig et al is assessed. The scores are compared for the 2 investigators as well as for the 3 investigation modes.
   4. Inclusion criteria

      * Age > 18 and < 80 years old
      * Given written informed consent
      * Patients with symptoms of deep venous thrombosis less than for 2 weeks
      * Thrombus occluding without any reperfusion in color mode in the common femoral vein (CFV), the femoral vein (FV) or the popliteal vein (PV)
   5. Exclusion criteria

      * Arterial occlusive disease
      * Acute myocardial infarction, symptoms of coronary artery disease
      * Pregnancy
      * History of stroke or transient ischemic attack
      * Arterial hypertension uncontrolled
      * Allergy to contrast media
      * Participation in another study
      * Right heart insufficiency (clinical assessment with jugular vein filling in 45° sitting position)
3. Study Endpoints

   Primary study endpoint:

   Detection of re - vascularization in > 3 months old thrombosis in patients with initially occluded veins, assessed with ultrasound contrast agent, the parameter used will be the difference between baseline and peak of the time intensity curve.

   Secondary study endpoint:

   Visibility of the newly developed small vessels in patients with occluding thrombus assessment during application of contrast agent, with color Doppler and power Doppler mode. The parameter used will be the visibility score.
4. Sample size

   Sample size is estimated to 9 patients in each group assuming a significant difference of 4.7 % for the mean values for the "time to peak" in patients with acute compared to chronic thrombosis with a significance level (alpha) of 0.05 and a power of 95 % (beta) assuming a standard deviation of 2. Sample size calculation was performed using Graphpad Prism 4.0b and StatMate 2.
5. Statistics

All parameters are analyzed as an independent unit. Statistical analysis will be calculated using the Stat View software package version 5.0 for Mac OS 9 (Stat View Software by Abacus C., Berkley, California) and Graph Pad Prism version 4 for Mac OS X (Graph Pad Software, San Diego, California). Results will be given in median and interquartile ranges. Comparison between visits in the same patients will be done by the non-parametric, paired Wilcoxon signed rank test or if more than two groups are involved the Kruskal Wallis test. A probability level of < 0.05 will be considered significant. The inter - reader agreement will be measured using the kappa value.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 80 years old
* Given written informed consent
* Patients with symptoms of deep venous thrombosis less than for 2 weeks Thrombus occluding without any reperfusion in color mode in the common femoral vein (CFV), the femoral vein (FV) or the popliteal vein (PV)

Exclusion Criteria:

* Arterial occlusive disease
* Acute myocardial infarction, symptoms of coronary artery disease
* Pregnancy
* History of stroke or transient ischemic attack
* Arterial hypertension uncontrolled
* Allergy to contrast media
* Participation in another study
* Right heart insufficiency (clinical assessment with jugular vein filling in 45° sitting position)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a newly diagnosed occluding venous thrombus with duplexsonography and symptoms of deep venous thrombosis less than for 2 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-07 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Vascularisation in thrombosis in patients with initially occluded veins, assessed with ultrasound contrast agent (relative difference between baseline and peak of the time intensity curve) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christina R. Jeanneret-Gris, MD, Principal Investigator — University of Freiburg
Locations (1):
- University of Freiburg, Freiburg im Breisgau, Baden Würtemberg, Germany